CLINICAL TRIAL: NCT00000718
Title: A Clinical Trial of Alternating and Intermittent Regimens of 2',3'-Dideoxycytidine and 3'-Azido-3'-Deoxythymidine in the Treatment of Patients With AIDS and Advanced ARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 047; 11021 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Dose-Response Relationship, Drug; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To determine if alternating zidovudine (AZT) and zalcitabine (dideoxycytidine; ddC) (first one and then the other) or intermittent therapy (1 week of drug then 1 week off) will lessen the toxic effects of either drug alone, while still inhibiting HIV (the AIDS virus) in patients with AIDS or AIDS related complex.

AZT extends the survival of some patients with AIDS, and both AZT and ddC are known to inhibit the growth of HIV. When AZT or ddC is given continuously over a prolonged period of time, toxic effects occur that are not found when the drugs are given for 4 - 6 weeks. It is hoped that by alternating the drugs or by giving one drug intermittently, the toxic effects can be decreased without lowering the therapeutic effectiveness of the drugs.

DETAILED DESCRIPTION:
AZT extends the survival of some patients with AIDS, and both AZT and ddC are known to inhibit the growth of HIV. When AZT or ddC is given continuously over a prolonged period of time, toxic effects occur that are not found when the drugs are given for 4 - 6 weeks. It is hoped that by alternating the drugs or by giving one drug intermittently, the toxic effects can be decreased without lowering the therapeutic effectiveness of the drugs.

Patients will be assigned to 1 of 7 treatment groups. Both AZT and ddC will be given by mouth every 4 hours. One group will take AZT continuously for 52 weeks. One group will alternate 1 week of AZT with a week with no drug for 48 weeks and another group will alternate 1 week of ddC with a week of no drug for 48 weeks. Other groups will alternate AZT and either low-dose or high-dose ddC on a weekly basis or a monthly basis for 48 weeks. Patients will be seen weekly for the first 8 weeks of study and less often thereafter. Blood samples will be withdrawn frequently and evaluated for possible changes in the immune system, toxic effects, and possible changes in the amount of HIV in the blood. Lumbar punctures and skin biopsies will also be performed.

AMENDED: All patients receiving continuous AZT will be switched to a lower dose of AZT if they have not already been switched. This is in accordance with results of NIAID ACTG 002, 016, and 019 which demonstrate that this dose of AZT delays progression of HIV symptoms.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Encouraged though not required:

* Inhaled pentamidine as prophylaxis for Pneumocystis carinii pneumonia (PCP).
* Allowed:
* AL-721 use is discouraged but not prohibited.
* Use of aspirin, acetaminophen, and nonsteroidal anti-inflammatory agents should be minimized, with continuous use for > 72 hours discouraged.
* Acute therapy (7 days) with oral acyclovir.
* Acute therapy with ketoconazole.

Concurrent Treatment:

Allowed:

* Up to 4 units of packed red blood cells for hemoglobin toxicity.

All patients must have the following:

* A consistently positive serum HIV p24 antigen = or > 70 pg/ml, defined by the Abbott HIV antigen test, on two occasions. The tests must be within 1 month of study entry, separated by at least 72 hours, and the last must be within 2 weeks of starting therapy. Any negative antigen test during the period will exclude the patient from the study.
* A positive antibody to HIV confirmed by any federally licensed ELISA test kit.
* Patients in group A must have AIDS related complex (ARC) as defined by the documented presence of at least one of the following:
* Recurrent oral candidiasis.
* Hairy leukoplakia.
* History of herpes zoster.
* Temperature > 38.5 degrees C with or without night sweats, persisting for > 14 consecutive days or > 15 days in a 30-day interval prior to study entry.
* Weight loss of > 15 lbs. or 10 percent of body weight noted in a 120-day period prior to study entry.
* Diarrhea defined as = or > 3 liquid stools per day, persisting for > 30 days prior to study entry without definable cause.
* Patients in group B must have CDC-defined AIDS not requiring systemic maintenance chemotherapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Transfusion dependence requiring 2 units of blood more than once per month.
* Significant malabsorption (> 10 percent weight loss within the past 3 months with serum carotene < 75 IU/ml or vitamin A < 74 IU/ml).
* Significant cardiac or liver disease.
* Significant neurologic abnormalities defined by any one of the following:
* A significant abnormality on the ddC Neuropathy Targeted Symptom Questionnaire defined as a symptom score > 4 (moderate severity) in any one of six categories or a score > 2 (mild severity) in any two of six categories.
* Moderate abnormalities on standardized neurologic exam.
* Any severe abnormality (a value = or > 4.0) on standardized 4-arm quantitative sensory testing of vibration threshold.
* Diabetes, renal failure, or alcoholism.
* Dose-limiting or transfusion-requiring toxicity during a previous course of zidovudine therapy.
* History of idiopathic thrombocytopenic purpura.
* Requirement for prolonged acyclovir therapy. Patients in group A must not have the following:
* Opportunistic infection or malignancy fulfilling the CDC definition of AIDS.
* Neoplasms other than basal cell carcinoma of the skin or in situ carcinoma of the cervix. Patients in group B must not have the following:
* Active opportunistic infection or AIDS-defining opportunistic infection requiring ongoing systemic therapy and/or prophylaxis other than inhaled pentamidine for Pneumocystis carinii pneumonia prophylaxis.
* Symptomatic visceral Kaposi's sarcoma (KS), progression of KS within the month prior to study entry.
* Concurrent neoplasms other than KS, basal cell carcinoma of the skin or in situ carcinoma of the cervix.

Concurrent Medication:

Excluded:

* Neurotoxic drugs.
* Prolonged acyclovir therapy.
* Antineoplastic therapy.
* Systemic therapy and/or prophylaxis for an AIDS-defining opportunistic infection, other than inhaled pentamidine for Pneumocystis carinii pneumonia (PCP) prophylaxis.
* Other antiretroviral agents, immunomodulators, or systemic corticosteroids.
* Other experimental medication.

Concurrent Treatment:

Excluded:

* Transfusion dependency (requiring 2 units of blood more than once per month).

Prior Medication:

Excluded:

* Antiretroviral agents within 60 days of study entry.
* Biologic modifiers or corticosteroids within 30 days prior to study entry.
* Dideoxycytidine (ddC).

Prior Treatment:

Excluded:

* Blood transfusion within 2 weeks of entry.

Any negative HIV p24 antigen test during the month prior to entry will exclude the patient from the study.

Active drug or alcohol abuse.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112
Dates: Study Completion 1991-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G Skowron, Study Chair
Locations (1):
- Northwestern University CRS, Chicago, Illinois, United States

REFERENCES:
- [Background] Lathey JL, Marschner IC, Kabat B, Spector SA. Deterioration of detectable human immunodeficiency virus serum p24 antigen in samples stored for batch testing. J Clin Microbiol. 1997 Mar;35(3):631-5. doi: 10.1128/jcm.35.3.631-635.1997. PMID 9041402
- [Background] Gries JM, Troconiz IF, Verotta D, Jacobson M, Sheiner LB. A pooled analysis of CD4 response to zidovudine and zalcitabine treatment in patients with AIDS and AIDS-related complex. Clin Pharmacol Ther. 1997 Jan;61(1):70-82. doi: 10.1016/S0009-9236(97)90183-1. PMID 9024175
- [Background] Merigan TC. Treatment of AIDS with combinations of antiretroviral agents. Am J Med. 1991 Apr 10;90(4A):8S-17S. doi: 10.1016/0002-9343(91)90405-m. PMID 1850192
- [Background] Skowron G, Merigan TC. Alternating and intermittent regimens of zidovudine (3'-azido-3'-deoxythymidine) and dideoxycytidine (2',3'-dideoxycytidine) in the treatment of patients with acquired immunodeficiency syndrome (AIDS) and AIDS-related complex. Am J Med. 1990 May 21;88(5B):20S-23S. doi: 10.1016/0002-9343(90)90417-c. PMID 2159705
- [Background] Skowron G, Bozzette SA, Lim L, Pettinelli CB, Schaumburg HH, Arezzo J, Fischl MA, Powderly WG, Gocke DJ, Richman DD, Pottage JC, Antoniskis D, McKinley GF, Hyslop NE, Ray G, Simon G, Reed N, LoFaro ML, Uttamchandani RB, Gelb LD, Sperber SJ, Murphy RL, Leedom JM, Grieco MH, Zachary J, Hirsch MS, Spector SA, Bigley J, Soo W, Merigan TC. Alternating and intermittent regimens of zidovudine and dideoxycytidine in patients with AIDS or AIDS-related complex. Ann Intern Med. 1993 Mar 1;118(5):321-30. doi: 10.7326/0003-4819-118-5-199303010-00001. PMID 8094279
- [Background] Fitzgibbon JE, Howell RM, Schwartzer TA, Gocke DJ, Dubin DT. In vivo prevalence of azidothymidine (AZT) resistance mutations in an AIDS patient before and after AZT therapy. AIDS Res Hum Retroviruses. 1991 Mar;7(3):265-9. doi: 10.1089/aid.1991.7.265. PMID 2064825